CLINICAL TRIAL: NCT01626066
Title: A Phase I Study of the Safety and Activation of a Cathepsin-Activatable Fluorescent Cancer Specific Probe LUM015
Brief Title: Cathepsin Activatable Fluorescent Probe
Acronym: LUM015
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Kirsch (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor-Investigator, David Kirsch, Associate Professor of Radiation Oncology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00035444
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoma; Soft Tissue Sarcoma; Breast Cancer
MeSH Terms: conditions — Sarcoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LUM015 (Experimental): Receive single dose of LUM015 through a vein in the arm the day prior to surgery
  Interventions: Drug: LUM015

INTERVENTIONS:
Drug: LUM015 — LUM015 assigned dose given once by IV push

SUMMARY:
Real-time detection of cancer cells during surgical removal of a tumor is important. Currently when tissue is removed at the time of surgery, the removed tissue goes to pathology when the margins (edges of the tissue) are examined to see if cancer cells are present. This may take a few to several days. Patients tissue with positive (cancer cells present) margins may require additional therapies including surgery. The purpose of this study is to determine a safe dose of a new imaging agent (LUM015), like a fluorescent contrast agent or dye, that will show in the tumor area during surgery and may help facilitate visualization of tumor for its removal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of soft tissue sarcoma and breast cancer patients scheduled for a lumpectomy or mastectomy.
* Subjects must be scheduled for surgical resection of a tumor at least 1 cm in size.
* Performance status of 0 or 1
* Able to read, understand and sign an informed consent form
* Must be able and willing to follow study procedures and instructions including a possible overnight stay before surgery
* Otherwise healthy except for the diagnosis of cancer
* ALT, AST, and total bilirubin within 1.5x institutional upper normal limits; and alkaline phosphatase within 2.5x institutional upper normal limits
* Serum creatinine of 1.5 mg or less; creatinine clearance greater than 30 ml/min
* May have previously received pre-operative external beam radiation therapy for this sarcoma

Exclusion Criteria:

* Pregnant or lactating
* Prolonged QT interval: corrected QT interval (QTc) > 480 msec
* Insulin dependent diabetes
* History of anaphylactic reactions to any drug or contrast agent
* Asthma under medical management
* Uncontrolled high blood pressure
* Severe, active co-morbidity
* Known substance addiction
* Sexually active and not willing/able to use medically acceptable forms of contraception.
* Obesity defined as BMI as body mass index greater than 35 kg/meter squared.
* Atopy or atopic syndrome
* Known AIDS
* Cannot have taken an investigational drug within 30 days of coming onto this study

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Dose of LUM015 in mg | 24 hours
  Dose of LUM015 in mg that is tolerated and labels tumors

SECONDARY OUTCOMES:
Mean number of fluorescence counts per second per square centimeter | At time of surgery
To obtain PK/PD information regarding LUM015 when administered IV in patients. | Two years
  The pharmacokinetic parameters to be measured will include: area under the curve (AUCt), maximum concentration (Cmax), time to maximum concentration (tmax) and first-order terminal (elimination) rate constant. Secondary (derived) parameters will include: terminal half-life (t1/2), clearance (CL), mean residence time (MRT), and apparent volume of distribution during the terminal phase (Vz). The distribution of these parameters will be described for each dose cohort separately; breast and sarcoma patients will be combined.
To analyze cathepsin protease expression in tumors. | 2 Years
  Cathepsin expression in tumors, measured in arbitrary units by Real-Time PCR compared to adjacent normal tissue when available, will be assessed in sarcomas and breast tumors. For each tissue specimen the expression of cathepsin will be compared to the imaging signal. Scatterplots of cathepsin level against imaging signal will be made according to tissue type within each dose cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Brigman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States